CLINICAL TRIAL: NCT02676609
Title: Assessment of the Impact of Food Carbohydrate and Insulin Dose Computing by an Application on Smart Phone on Glucose Control in Patients With Type 1 Diabetes
Brief Title: Impact of Food Carbohydrate and Insulin Dose Computing by on Smart Phone on Glucose Control in Patients With Diabetes
Acronym: GLUCAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Université Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: UF 9665
Record Dates: First submitted 2016-02-03; First posted 2016-02-08 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Smart phone application; carbohydrate counting; meal insulin dose
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Use of smart phone application (device glucal) (Active Comparator): Before each meal patient will enter in the application food intakes. Automated carbohydrate and meal insulin dose computing according to individual meal insulin/carbohydrate ratio.
  During the first month, then during the second month they'll use as usual their traintement and meal without the apllication
  Interventions: Device: Automated carbohydrate and meal insulin dose computing
- Use of smart phone application (second month) (Active Comparator): During the first month they'll use as usual their traintement and meal without the apllication ,then during the second month they'll use the apllicatioin.
  Before each meal patient will enter in the application food intakes. Automated carbohydrate and meal insulin dose computing according to individual meal insulin/carbohydrate ratio.
  Interventions: Device: Automated carbohydrate and meal insulin dose computing

INTERVENTIONS:
Device: Automated carbohydrate and meal insulin dose computing — Use of smart phone application will compute carbohydrate amount and meal insulin dose according to individual meal insulin/carbohydrate ratio.

SUMMARY:
During this study, we will assess a new smart phone application which aims at helping patients with Type 1 diabetes to compute food carbohydrates and meal insulin doses. Patients, already trained to carbohydrate counting, will be recruited among those who have been using this method daily for at least 6 months. They will complete two one-month study phases, using the application in one phase and counting carbohydrate and insulin doses without the application in the other phase, with randomized order of each phase. Visits are scheduled at the start and at the end of each phase to collect data on glucose control and insulin doses. Questionnaires assessing health-related quality of life and ability of self-management of diabetes will also be filled by patients before and after each study phase.

DETAILED DESCRIPTION:
During this study, we will assess a new smart phone application which aims at helping patients with Type 1 diabetes to compute food carbohydrates and meal insulin doses. Patients, already trained to carbohydrate counting, will be recruited among those who have been using this method daily for at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes since more than 1 year
* Basal-bolus insulin regimen since more than 6 months
* Daily practice of food carbohydrate counting since more than 6 months
* HbA1c level below 12%

Exclusion Criteria:

* Type 2 diabetes
* No ability to use a smart phone
* Pregnancy or lactation
* Severe psychiatric disorders
* Eating disorders
* Alcohol abuse or recreational drug use

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
2-hour postmeal blood glucose values between 80 and 180 mg/dl | 4 weeks
  Percent 2-hour postmeal blood glucose values between 80 and 180 mg/dl during 4 weeks

SECONDARY OUTCOMES:
Mean 2-hour postmeal blood glucose level | 4 weeeks
  Average 2-hour postmeal blood glucose level during 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eric Renard, MD, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Hôpital Lapeyronie, Montpellier, Hérault, France

IPD SHARING:
Plan to Share IPD: Undecided